CLINICAL TRIAL: NCT03565263
Title: Functional Gastrointestinal Disorders in Children and Adolescents With Inflammatory Bowel Disease in Remission: Prevalence and Identification of Clinical and Psychosocial Risk Factors
Brief Title: Functional Gastrointestinal Disorders in Pediatric IBD
Acronym: TFI-MICI
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-160
Record Dates: First submitted 2018-02-09; First posted 2018-06-21 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Inflammatory Bowel Diseases; Functional Gastrointestinal Disorders; Pediatric Disorder; Anxiety Depression; Quality of Life
MeSH Terms: conditions — Inflammatory Bowel Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FGID-IBD: * Patients aged 9-18 years
  * with inflammatory bowel disease (Crohns, ulcerative colitis or indeterminate colitis)
  * in remission (defined as: Physician's global assessment = remission, no nocturnal stools, no blood in stools, < or = 3 stools/day, C-reactive-protein < 10 mg/L, Erythrocyte sedimentation rate < 20 mm, no flare of disease or change of treatment in the last 3 months, no ongoing corticosteroid therapy
  * followed for IBD for at least 1 year
  * with at least one Functional Gastrointestinal disorder according to the Fr-qPGS questionnaire (Rome III criteria)
- No FGID-IBD: * Patients aged 9-18 years
  * with inflammatory bowel disease (Crohns, ulcerative colitis or indeterminate colitis)
  * in remission (defined as: Physician's global assessment = remission, no nocturnal stools, no blood in stools, < or = 3 stools/day, C-reactive-protein < 10 mg/L, Erythrocyte sedimentation rate < 20 mm, no flare of disease or change of treatment in the last 3 months, no ongoing corticosteroid therapy
  * followed for IBD for at least 1 year
  * not a single Functional Gastrointestinal disorder according to the Fr-qPGS questionnaire (Rome III criteria)

SUMMARY:
Background: Persistent gastrointestinal symptoms have been described in patients who are considered in remission of their inflammatory bowel disease (IBD). These symptoms, attributed to Functional gastrointestinal disorders (FGID) in IBD, may have a significant impact of quality of life, and may be associated with fatigue, anxiety and depression. There is very little data regarding pediatric specificities of these FGID.

Aims: The aim of the study is to evaluate the prevalence of FGID in pediatric patients with IBD in remission. Secondary aims are to investigate a possible association of FGID with fatigue, anxiety, depression and impacted quality of life in the patients, as well as anxiety and depression in the parents.

Methods: This will be an observational, case-control study. All patients between 9 and 18 years old , with IBD in remission will be invited to participate. Questionnaires will be web-based and will evaluate: presence of FGID (Fr-qPGS), fatigue (FACIT-F), anxiety (SCARED-R), depression (CDI), quality of life (IMPACT-III). Parents will be invited to fill in web-based questionnaires on their symptoms of anxiety (STAI/Y-A and STAI/Y-B) and depression (BDI). Clinical parameters will be retrieved retrospectively from the chart. Level of remission will be confirmed by most recent blood tests and fecal calprotectin. Patients with FGID will be compared to patients without FGID in terms of clinical characteristics, disease phenotype and associated psychological comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* IBD (Crohns disease, Ulcerative colitis or IBD-U)
* in remission (defined as: Physician's global assessment = remission, no nocturnal stools, no blood in stools, < or = 3 stools/day, C reactive protein < 10 mg/L, erythrocyte sedimentation rate < 20 mm, no flare of disease or change of treatment in the last 3 months, no ongoing corticosteroid therapy
* followed for IBD for at least 1 year

Exclusion Criteria:

* presence of an ileostomy or colostomy
* past history of total colectomy
* unable to understand written French or to answer the questionnaires

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In the aim of recruiting a sample that will be the most representative possible of the population of pediatric IBD patients in remission in France, patients will be recruited for the study through different procedures:
  * either during a routine visit to the pediatric gastroenterology clinic (all French pediatric gastroenterology clinics will be study centers)
  * or during a routine visit to the adult gastroenterology clinic (the French adult gastroenterologists will be informed of the study and will be able to apply to be a study center)
  * finally, the patient will be able to find information on the study through the French IBD patient Foundation (association Francois Aupetit) and contact the investigators in order to participate.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2020-11-08 (Actual)

PRIMARY OUTCOMES:
Presence of Functional Gastrointestinal Disorder | baseline
  Rome III criteria for FGID (Fr-qPGS questionnaire)

SECONDARY OUTCOMES:
Anxiety | baseline
  SCARED-R questionnaire
Depression | baseline
  CDI questionnaire
Quality of life - disease related | baseline
  IMPACT-III questionnaire
Fatigue | baseline
  peds FACIT-F questionnaire
Anxiety (parents) | baseline
  STAI/Y-A and STAI/Y-B questionnaires
Depression (parents) | baseline
  BDI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claire Dupont-Lucas, Principal Investigator — Groupe d'Etudes Therapeutiques des Affections Inflammatoires Digestives pediatriques
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No